CLINICAL TRIAL: NCT01345812
Title: Time-lapse Assessed Evaluation of Embryo Development After Stimulation With Either Recombinant Follicle Stimulating Hormone (FSH) or Urine-derived Follicle Stimulating Hormone (FSH).
Brief Title: Time-lapse Evaluation of Embryo Development After Stimulation With One of Two Different Gonadotrophins.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of patients for recruitment
Sponsor: University of Aarhus (Other)
Collaborators: The Fertility Clinic Braedstrup Hospital (Unknown); Herlev Hospital (Other); Odense University Hospital (Other); Trianglen Fertility Clinic (Unknown); Aagaard Fertility Clinic (Other); Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20090169
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Patients for In Vitro Fertilization(IVF)Treatment
Keywords: ART; IVF; Timelapse
MeSH Terms: interventions — follitropin alfa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- urine-derived FSH (Active Comparator): Follicle stimulating hormone
  Interventions: Drug: HP-HMG
- recombinant FSH (Active Comparator): Follicle stimulation hormone
  Interventions: Drug: recombinant FSH

INTERVENTIONS:
Drug: HP-HMG — 100 - 300 IU for stimulation of women in ART treatment
  Other Names: Menopure
  Arms: urine-derived FSH
Drug: recombinant FSH — 100 -300 IU for stimulation of women in ART treatment
  Other Names: Gonal-F
  Arms: recombinant FSH

SUMMARY:
The primary purpose of the investigation is to identify differences in embryo development after follicle stimulation with two different gonadotrophins.

DETAILED DESCRIPTION:
So far the assessment of the development potential of the single embryo has been limited by the vulnerability of the embryos when exposed to fluctuations in temperature and CO2 levels.

Thus embryos can only be allowed to leave incubators for a very limited time period.

However, with the development of time-lapse systems for clinical use it is possible to make continuous time-lapse recordings of embryos while they are in a safe incubator environment.

The embryos are not compromised, but the entire embryonic development can still be seen, and will subsequently provide new and essential information on the competence of the single embryo.

Based on the above it is expected that the probability of selecting the most viable and competent embryo is increased, which, in turn, will increase the success rate for couples seeking infertility treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants(heterosexuals, lesbian couples and single women) must sign a document of informed consent

* Female age 21-45 years(both inclusive)
* Patients for IVF treatment
* Regular menstrual cycle 21-35 days(both inclusive)
* Normal FSH levels(1-15 IU/L)
* BMI between 18-32(both inclusive)
* Patients must be able to read and understand patient information in national language

Exclusion Criteria:

PCO

- Endometriosis as primary diagnosis

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 291 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of Top Quality Embryos day 2 | 44 h after insemination
  The oocytes are inseminated and loaded to the time-lapse instrument and cultured for two days. The embryo developemnt are followed at the movie and the embryos are scored according to a standard scoring criteria at 44 h after insemination

SECONDARY OUTCOMES:
Implantation rate | 5 weeks after embryo transfer
  The pregnancy is verified by a blood sample two weeks after embryo transfer and the number of embryos implanted are verified by ultrasound scanning five weeks after embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Inge Agerholm, Phd, Principal Investigator — IVF clinic Braedstrup
Locations (1):
- The fertility clinic, Brædstrup, Denmark

REFERENCES:
- See also: database — http://www.ncbi.nlm.nih.gov/pubmed/